CLINICAL TRIAL: NCT03399708
Title: Immune Metabolic Associations in Psoriatic Arthritis Study
Brief Title: Immune Metabolic Associations in Psoriatic Arthritis
Acronym: IMAPA
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN16RH008
Record Dates: First submitted 2017-11-27; First posted 2018-01-16 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Psoriasis; Psoriatic Arthritis
Keywords: apremilast; PDE4 inhibition; cardiometabolic; immune profile
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — apremilast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Routine blood (FBC, creatinine and/or GFR, LFTs) Acute phase reactants: ESR, CRP Oral Glucose Tolerance test (OGTT) = 0,30,60,90,120min (glucose, insulin) =0, 30, 120 min (GLP-1) Fasting lipids, HbA1c, glucose, insulin, GLP-1 levels Blood samples for NMR metabolomic profiling Circulating cytokines & adipokines
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Apremilast 30mg — Apremilast will used in line with its license. This includes the standard dose titration scheme (see section 6) and then the usual maintenance dose of 30 mg twice daily orally.

SUMMARY:
To use apremilast in clinical practice as a molecular probe to evaluate the effects of PDE4 inhibition on the cardiometabolic status and immune profile in patients with PsA and psoriasis.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) and psoriasis are characterised by immune, metabolic, and vascular dysfunction. There is an increase in Major Adverse Cardiovascular Events in people with PsA and psoriasis not explained by conventional cardiovascular risk factors. Furthermore, obesity in psoriasis is associated with increased risk of developing PsA3. Dietary interventions leading to weight loss >5% are associated with a higher rate of achievement of minimal disease activity in overweight/obese patients with PsA treated with TNF inhibitors. Phosphodiesterase 4 (PDE4) inhibition with apremilast is licensed for the treatment of PsA and psoriasis and has been noted to be associated with weight loss. There is also data from animal models to suggest a role for PDE4 in glucose metabolism. However, the exact mechanisms underlying this are unclear and warrant investigation in humans. PDE4 may help explain the link between the immune and cardiometabolic dysfunction that characterises PsA and psoriasis, with pathogenic and therapeutic implications.

This study aims to use apremilast as a clinical molecular probe to evaluate the effects of PDE4 inhibition on metabolic, vascular, and immune status in patients with PsA and psoriasis. The hypothesis is that PDE4 inhibition mediates profound and synergistic effects on immune and metabolic pathways in these conditions to improve metabolic status and normalise dysregulated immunity.

Measurement of metabolic, immunological and vascular outcomes in 60 patients (40 with PsA and 20 with psoriasis) receiving apremilast as part of their standard clinical care will be taken. A subgroup of 20 participants with PsA will also undergo more in-depth investigations including MRI of abdominal fat, subcutaneous fat biopsy, measurement of vascular endothelial function using EndoPAT and more detailed deep-immunophenotyping. Patients will be recruited from rheumatology and dermatology clinics in NHS Greater Glasgow and Clyde (primary site) and two other recruiting sites in Scotland via the Scottish Collaborative Arthritis Research network (SCAR).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Have either a diagnosis of PsA (n=40) fulfilling the CASPAR criteria or Chronic plaque psoriasis (confirmed by dermatologist) (n=20)
3. Eligible for apremilast therapy in line with the licence and SMC approval
4. Able and willing to give written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

1. History of or current autoimmune rheumatic disease other than PsA or psoriasis
2. Severe renal disease (eGFR ≤30ml/min)
3. Liver disease with ALT/AST >4 times ULN
4. Haemoglobin ≤9 g/dl
5. Inflammatory bowel disease or coeliac disease
6. Patients with any cancer currently receiving chemo- or radiotherapy
7. Severe depression and/or history of suicidal ideation or attempts.
8. Currently receiving other leflunomide or biologics
9. Current oral steroids or IM steroids within 6 weeks of baseline.
10. Clinically meanigful weight loss of >3kg, current or planned use of weight loss medication e.g. orlistat, or severe calorie restriction within the first 3 months of the study
11. Current insulin therapy for diabetes
12. Current use of GLP-1 agonists or dipeptidyl peptidase-4 (DPP-IV) inhibitors
13. Statin therapy started/stopped or dose altered within 3 months of baseline visit
14. Thyroxine started or dose altered within 6 weeks of baseline
15. Acitretin within 8 weeks of baseline
16. Pregnancy or breast feeding
17. Women planning to become pregnant during the study period
18. Women of reproductive age or male partners of women of reproductive age unwilling to use effective contraception while taking apremilast & for at least 28 days after last dose of apremilast
19. Known HIV, hepatitis B and C infection
20. Patient unable to participate in long term data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PsA and psoriasis.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-10-12 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Changes in cardiometabolic profile | 3 months
  To characterise dynamic changes in cardiometabolic profile with formal assessment at 3 months.

SECONDARY OUTCOMES:
Lipids | 6 months
  Change in lipid profile
NMR metabolomic profile | 6 months
  Change in NMR metabolomic profile
Blood pressure | 6 months
  Change in blood pressure
endothelial function | 3 months
  change in endothelial function
MRI imaging | 3 months
  change in visceral, subcutaneous, liver, and pancreatic fat as assessed by MRI imaging
GLP-1 levels | 6 months
  Change in fasting & post-prandial GLP-1 levels
adipose tissue | 3 months
  Change in adipose tissue composition
immune profile | 6 months
  Change circulating cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Siebert, MBChB PhD, Principal Investigator — Glasgow University and NHS GGC
Locations (1):
- Glasgow Royal Infirmary, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided